CLINICAL TRIAL: NCT01499771
Title: A Bioequivalence Study Of 80 Mg Atorvastatin Calcium Tablets Versus 80 Mg Lipitor® Tablets Under Fed Conditions.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R09-1033
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Atorvastatin Calcium Tablets of OHM Laboratories Inc.
  Interventions: Drug: Atorvastatin
- 2 (Active Comparator): LIPITOR® Tablets 80mg of Pfizer Ireland Pharmaceuticals
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 80 Mg tablets

SUMMARY:
This study assessed the relative bioavailability of 80 mg Atorvastatin Calcium Tablets (containing atorvastatin calcium equivalent to 80 mg atorvastatin) manufactured by OHM Laboratories, Inc., USA (A subsidiary of Ranbaxy Pharmaceuticals., USA) compared to that of 80 mg LIPITOR® Tablets (containing atorvastatin calcium equivalent to 80 mg atorvastatin) distributed by Parke Davis, Division of Pfizer Inc., USA following a single oral dose (1 x 80 mg tablet) in healthy adult subjects when administered under fed conditions.

DETAILED DESCRIPTION:
This was an open-label, balanced, randomized, two-period, two-treatment, two-sequence, single-dose crossover bioequivalence study under fed conditions. The total duration of the study, screening through study exit, was approximately 8 weeks with at least a 14-day washout period between doses. At study check-in, the subjects reported to the clinical site at least 36 hours prior to Day 1 dosing and were required to stay for 24 hours after Day 1 dosing. Blood sample collections were obtained within 90 minutes prior to dosing (0 hour) and after dose administration at 0.333, 0.667, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60, 72, and 96 hours. A total of 25 blood samples were collected per study period for a total of 50 samples or 150 mL total volume.

ELIGIBILITY:
Inclusion Criteria:

1. Informed of the nature of the study, had agreed to, and was able to read, review, and sign the informed consent document prior to Period I dosing. The informed consent document was written in English, therefore the volunteer must have had the ability to read and communicate in English.
2. Completed the screening process within four weeks prior to Period I dosing.
3. Healthy male or female, 18 years of age or older at the time of dosing.
4. Body mass index (BMI) between 18 - 32 kg/m2, inclusive, and weighed at least 110 lbs.
5. Generally healthy as documented by medical history, physical examination (including but not limited to an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems), vital sign assessments, 12-lead ECG, clinical laboratory assessments, and by general observations. Any abnormalities/deviations from the acceptable range that might have been considered clinically relevant by the study physician or investigator were evaluated as individual cases, documented in study files, and agreed upon by the principal investigator (or sub-investigator) prior to enrolling the subject in this study.
6. Female subjects were:

   * of postmenopausal status (no menses) for at least one year and if < 55 years of age had documented FSH level ≥ 40 mIU/mL; or,
   * sterile [surgically (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or the Essure® Procedure].

Fe Female subjects that were surgically sterile were to provide documentation of the bilateral tubal ligation, bilateral oophorectomy, or hysterectomy prior to Period I dosing. The Essure® Procedure must have been inserted at least 3 months prior with documentation of the Essure® confirmation test prior to Period I dosing.

Exclusion Criteria:

1. Reported receiving any investigational drug within 28 days prior to Period I dosing.
2. Reported any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the clinical investigator(s).
3. Clinical laboratory test values outside the accepted range and when confirmed on re-examination was deemed to be clinically significant.
4. When confirmed upon additional testing, demonstrates a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
5. Reported a clinically significant illness during the 28 days prior to Period I dosing (as determined by the clinical investigators).
6. Demonstrated a positive drug screen or alcohol breath test.
7. Reported a history of allergic response(s) to atorvastatin or related drugs.
8. Reported a history of clinically significant allergies including food or drug allergies.
9. Reported a history of drug or alcohol addiction or abuse within the past year.
10. Reported donating blood within 28 days prior to Period I dosing. All subjects were to be advised not to donate blood for four weeks after completing the study.
11. Reported donating plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects were to be advised not to donate plasma for four 12. weeks after completing the study.

13. Reported an intolerance of direct venipuncture. 14. Reported difficulty fasting or consuming standardized meals. 15. Reported difficulty swallowing tables or capsules whole. 16. Pregnant, lactating, breastfeeding, or intended to become pregnant over the course of the study (females only).

17. Demonstrates a positive pregnancy screen (female only).

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Atorvastatin. | 0, 0.333, 0.667, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 6, 8, 10, 12, 16, 24, 36, 48, 60, 72, and 96 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Research 4801 Amber Valley Parkway, Fargo, North Dakota, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html